CLINICAL TRIAL: NCT00600223
Title: Functional Voice and Speech Outcomes Following Surgical Voice Restorations: A Comparison of Pharyngeal Reconstruction Approaches
Brief Title: Functional Voice and Speech Outcomes Following Surgical Voice Restorations: A Comparison of Pharyngeal Construction Approaches
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Massachusetts Eye and Ear Infirmary (Other); Brigham and Women's Hospital (Other)
Responsible Party: Dennis Kraus, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 05-104
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-10

CONDITIONS: Larynx Cancer
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients undergoing laryngectomy and pharyngeal reconstruction
  Interventions: Behavioral: questionnaires and standardized, digital voice recording

INTERVENTIONS:
Behavioral: questionnaires and standardized, digital voice recording — Patient will be asked to complete four sets of forms. Upon completion of these forms, the study subject and the investigator will proceed to a quiet room for the standardized, digital voice recording. Recording will be made on digital audiotape using a standardized portable, digital audio recorder.

SUMMARY:
The purpose of this study is to evaluate the nature and quality of speech after removal of the voice box and all or part of the swallowing tube.

The study is evaluating which type of surgery provides patients with the best speech and voice.

These data will be used to help surgeons to design better ways to restore voice function after removal of the voice box. Information about disease, its treatment, quality of life, and physical and vocal function will be collected. An audio recording of vocal tasks will also be done. All of this information will be analyzed and the two different subject groups will be compared to see if there are differences.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have undergone removal of the larynx and the entire pharynx by either traditional reconstruction or more advanced reconstructive techniques, which involve the use of tissue, such as skin or bowel, from other parts of the body. There is no time frame for reconstruction. All subjects who have previously undergone reconstruction are eligible.
* Subjects who use the tracheoesophageal puncture method of voice restoration as their primary communication technique.
* > or equal to 18 years old

Exclusion Criteria:

* Do not have functional voice restoration.
* Do not speak English as a functional language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinic
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2005-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Determine the pertinent differences in objective and subjective voice parameters between PR techniques, specifically comparing those techniques that provide mucosal lining (jejunum) to those with cutaneous lining (radial forearm flap). | conclusion of study

SECONDARY OUTCOMES:
Provide physician with meaningful and relevant data upon which to base the optimal choice of pharyngeal reconstruction method for individual patients who must undergo laryngectomy with pharyngeal reconstruction for the treatment of carcinoma. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Kraus, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org